CLINICAL TRIAL: NCT04371016
Title: Pulmonary and Ventilatory Effects of Bed Verticalization in Patients With Acute Respiratory Distress Syndrome: An Exploratory and Pathophysiology Study
Brief Title: Pulmonary and Ventilatory Effects of Bed Verticalization in Patients With Acute Respiratory Distress Syndrome
Acronym: ERECTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP AUDARD 2019
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Mechanical Ventilation; Verticalization; Intensive Care Unit
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Beds

STUDY DESIGN:
Intervention Model Description: Interventional study evaluating the beneficial impact of verticalization of patients with ARDS on pathophysiological parameters
Masking Description: Analysis of data will be conducted by a statistician not involved in interventions at bedside
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verticalization group (Experimental): After checking the availability of the bed dedicated to verticalization (Total Lift Bed™, VitalGo Systems, Inc., Arjo AB), the inclusion and non-inclusion criteria, as well as the morphology of lung injury, the patient is included. The following procedures are performed :
  * insertion of an esophageal balloon catheter (Nutrivent®, Sidam)
  * installation of an EIT belt in the 4th or 5th intercostal space (Pulmovista® 500, Dräger)
  * insertion of a Swan-Ganz catheter
  * continuous recording of digital and analogic data
  After collecting initial data from the patient in a strict lying position at 0°, successive 30-minutes position steps at 30°, 60° and 90° will be performed. At the end of the 30 minutes, and for each step, all the data is collected.
  Interventions: Other: Verticalization (bed)

INTERVENTIONS:
Other: Verticalization (bed) — The use of a dedicated bed (Total Lift Bed™, VitalGo Systems, Inc., Arjo AB) allows the verticalization of patients under sedation and mechanical ventilation up to 90°. The procedure foresees the gradual verticalization of the patients of 0°, 30°, 60° and 90° by steps of 30 minutes.
  At the end of each position step (0°, 30°, 60° and 90°), measurement of end-expiratory lung impedance (EELI) and chest electrical impedance tomography (EIT) parameters, measurement of esophageal pressures, collection of ventilatory parameters on the ventilator, collection of Swan-Ganz catheter hemodynamic data, measurement of lung shunt by mixed venous and arterial blood gas analyses and measurement of end-expiratory lung volume (EELV) by the N2 washin-washout method

SUMMARY:
Acute respiratory distress syndrome (ARDS) is defined using the clinical criteria of bilateral pulmonary opacities on a chest radiograph, arterial hypoxemia (partial pressure of arterial oxygen [PaO2] to fraction of inspired oxygen [FiO2] ratio ≤ 300 mmHg with positive end-expiratory pressure [PEEP] ≥ 5 cmH2O) within one week of a clinical insult or new or worsening respiratory symptoms, and the exclusion of cardiac failure as the primary cause. ARDS is a fatal condition for intensive care unit (ICU) patients with a mortality between 30 and 40%, and a frequently under-recognized challenge for clinicians. Patients with severe symptoms may retain sequelae that have recently been reported in the literature. These sequelae may include chronic respiratory failure, disabling neuro-muscular disorders, and post-traumatic stress disorder identical to that observed in soldiers returning from war.

The management of a patient with ARDS requires first of all an optimization of oxygenation, which relies primarily on mechanical ventilation, whether invasive or non-invasive (for less severe patients). Since the ARDS network study published in 2000 in the New England Journal of Medicine, it has been internationally accepted that tidal volumes must be reduced in order to limit the risk of alveolar over-distension and ventilator-induced lung injury (VILI). A tidal volume of approximately 6 mL.kg-1 ideal body weight (IBW) should be applied. Routine neuromuscular blockade of the most severe patients (PaO2/FiO2 < 120 mmHg) is usually the rule, although it is increasingly being questioned. Comprehensive ventilatory management is based on the concepts of baby lung and open lung, introduced respectively by Gattinoni and Lachmann. According to these concepts, it must be considered that the lung volume available for mechanical ventilation is very small compared to the healthy lung for a given patient (baby lung) and that the reduction in tidal volume must be associated with the use of sufficient PEEP and alveolar recruitment maneuvers to keep the lung "open" and limit the formation of atelectasis.

In addition to this optimization of mechanical ventilation, it is possible to reduce the impact of mechanical stress on the lung. The prone position, for example, makes it possible to free from certain visceral and mediastinal constraints, to optimize the distribution of ventilation as well as the ventilation to perfusion ratios.

Thanks to the technological progress of intensive care beds, it is now possible to verticalize ventilated and sedated patients in complete safety. Verticalization could reduce the constraints imposed to the lungs, by reproducing the more physiological vertical station, and thus modifying the distribution of ventilation.

Indeed, in two physiological studies published in 2006 and 2013 in Intensive Care Medicine, 30 to 40% of patients with ARDS appeared to respond to partial body verticalization at 45° and 60° (in a semi-seated or seated position). In addition to improving arterial oxygenation, verticalization appeared to decrease ventilatory stress, related to supine position, and increase alveolar recruitment, with improved lung compliance and end-expiratory lung volume (EELV) over time. Nevertheless, 90° verticalization has never been studied, nor have positions without body flexion (seated or semi-seated). In these studies, only patients with the highest lung compliance appeared to respond. These data support the current hypothesis of subgroups of patients with ARDS with different pathophysiological characteristics (morphological and phenotypic) and therapeutic responses.

The investigators hypothesize that verticalization of patients with ARDS improves ventilatory mechanics by reducing the constraints imposed on the lung (transpulmonary pressure), pulmonary aeration, arterial oxygenation and ventilatory parameters.

The first objective is to study the influence of the bed position of the patient with early ARDS on the variations in respiratory mechanics represented by the transpulmonary driving pressure (ΔPtp). The second objective is to evaluate changes in ventilatory physiology, tolerance and feasibility of verticalization in patients with early ARDS.

DETAILED DESCRIPTION:
This is an interventional study evaluating the beneficial impact of verticalization of patients with ARDS on pathophysiological parameters.

This therapeutic study aims to test patient's position using dedicated beds (Total Lift Bed™, VitalGo Systems Inc., Arjo AB). The study consists of comparing pulmonary pathophysiological parameters for different positions (from the strict dorsal decubitus to the vertical, with 30° and 60° steps) in patients with early ARDS of focal and non-focal morphologies, under invasive mechanical ventilation.

The primary outcome is the difference between the transpulmonary driving pressure (ΔPtp) measured at the end of each verticalization step (30th minute) and the basal value measured at the beginning of the protocol, in strict dorsal decubitus (0°).

The minimum number of subjects to enroll in this study is 30 patients with early ARDS, including 15 with focal lung morphology and 15 with non-focal lung morphology. Intermediate analyses are planned every 5 patients in order to reevaluate the needed number of patients.

The use of a dedicated bed (Total Lift Bed™, VitalGo Systems, Inc., Arjo AB) allows the verticalization of patients under sedation and mechanical ventilation up to 90°. The procedure foresees the gradual verticalization of the patients of 0°, 30°, 60° and 90° by steps of 30 minutes. At the end of each position step (0°, 30°, 60° and 90°), measurement of end-expiratory lung impedance (EELI) and chest electrical impedance tomography (EIT) parameters, measurement of esophageal pressures, collection of ventilatory parameters on the ventilator, collection of Swan-Ganz catheter hemodynamic data, measurement of lung shunt by mixed venous and arterial blood gas analyses and measurement of end-expiratory lung volume (EELV) by the N2 washin-washout method.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate or severe Acute Respiratory Distress Syndrome (ARDS) (PaO2/FiO2 < 200 mmHg), at their early phase (< 12h), under invasive mechanical ventilation with controlled ventilation (intubation or tracheotomy).
* Patient equipped with an arterial catheter.
* Patient sedated (BIS between 30 and 50) and, if necessary, under neuromuscular blocking agent (TOF < 2/4 at the orbicular) to avoid inspiratory effort.
* Patient hemodynamically optimized following the Swan-Ganz catheter data.

Exclusion Criteria:

* Refusal to participate in the proposed study.
* Unavailability of the bed dedicated to verticalization (Total Lift Bed™, VitalGo Systems Inc., Arjo AB)
* Obesity with BMI ≥ 35 kg.m-2
* Significant hemodynamic instability defined as an increase of more than 20% in catecholamine doses in the last hour, despite optimization of blood volume, for a target mean blood pressure between 65 and 75 mmHg.
* Contraindication to the insertion of a nasogastric tube
* Contraindication to the use of the chest electrical impedance tomography
* Contraindication to the insertion of a Swan-Ganz catheter
* Contraindication to the application of compression stockings
* Patient under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Transpulmonary driving pressure (ΔPtp) | At the end of each verticalization step (30th minute)
  Difference between the transpulmonary driving pressure (ΔPtp) measured at the end of each verticalization step (30th minute) and the basal value measured at the beginning of the protocol, in strict dorsal decubitus (0°).

SECONDARY OUTCOMES:
Pulmonary mechanics | Baseline
  Maximal transpulmonary pressure (alveolar stress)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Maximal transpulmonary pressure (alveolar stress)
Pulmonary mechanics | Baseline
  Alveolar strain (Vt/EELV)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Alveolar strain (Vt/EELV)
Pulmonary mechanics | Baseline
  Driving pressure
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Driving pressure
Pulmonary mechanics | Baseline
  Transpulmonary driving pressure
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Transpulmonary driving pressure
Pulmonary mechanics | Baseline
  Dead space (Vd/Vt)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Dead space (Vd/Vt)
Pulmonary mechanics | Baseline
  Pulmonary compliance
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Pulmonary compliance
Pulmonary mechanics | Baseline
  Pressure-volume curves
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Pressure-volume curves
Pulmonary mechanics | Baseline
  Recruitable volume
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Recruitable volume
Pulmonary mechanics | Baseline
  Optimal PEEP (best compliance)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Optimal PEEP (best compliance)
Pulmonary mechanics | Baseline
  O2 consumption (VO2)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  O2 consumption (VO2)
Pulmonary mechanics | Baseline
  CO2 production (VCO2)
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  CO2 production (VCO2)
Pulmonary mechanics | Baseline
  Pulmonary shunt
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Pulmonary shunt
Pulmonary mechanics | Baseline
  Mechanical power imparted to patient's lungs by ventilator
Pulmonary mechanics | At the end of each verticalization step (30th minute)
  Mechanical power imparted to patient's lungs by ventilator
Chest electrical impedance tomography (EIT) | Baseline
  Center Of Ventilation (COV)
Chest electrical impedance tomography (EIT) | At the end of each verticalization step (30th minute)
  Center Of Ventilation (COV)
Chest electrical impedance tomography (EIT) | Baseline
  Tidal Impedance Variation (TIV)
Chest electrical impedance tomography (EIT) | At the end of each verticalization step (30th minute)
  Tidal Impedance Variation (TIV)
Chest electrical impedance tomography (EIT) | Baseline
  Regional Ventilation Delay (RVD)
Chest electrical impedance tomography (EIT) | At the end of each verticalization step (30th minute)
  Regional Ventilation Delay (RVD)
Chest electrical impedance tomography (EIT) | Baseline
  End Expiratory Lung Impedance (EELI)
Chest electrical impedance tomography (EIT) | At the end of each verticalization step (30th minute)
  End Expiratory Lung Impedance (EELI)
Chest electrical impedance tomography (EIT) | Baseline
  Percentages of over-distended and collapsed alveolar regions.
Chest electrical impedance tomography (EIT) | At the end of each verticalization step (30th minute)
  Percentages of over-distended and collapsed alveolar regions.
Hemodynamics | Baseline
  Heart rate
Hemodynamics | At the end of each verticalization step (30th minute)
  Heart rate
Hemodynamics | Baseline
  Invasive systolic blood pressure
Hemodynamics | At the end of each verticalization step (30th minute)
  Invasive systolic blood pressure
Hemodynamics | Baseline
  Invasive mean blood pressure
Hemodynamics | At the end of each verticalization step (30th minute)
  Invasive mean blood pressure
Hemodynamics | Baseline
  Invasive diastolic blood pressure
Hemodynamics | At the end of each verticalization step (30th minute)
  Invasive diastolic blood pressure
Hemodynamics | Baseline
  Continuous cardiac output
Hemodynamics | At the end of each verticalization step (30th minute)
  Continuous cardiac output
Hemodynamics | Baseline
  Pulmonary systolic arterial pressures
Hemodynamics | At the end of each verticalization step (30th minute)
  Pulmonary systolic arterial pressures
Hemodynamics | Baseline
  Pulmonary mean arterial pressures
Hemodynamics | At the end of each verticalization step (30th minute)
  Pulmonary mean arterial pressures
Hemodynamics | Baseline
  Pulmonary diastolic arterial pressures
Hemodynamics | At the end of each verticalization step (30th minute)
  Pulmonary diastolic arterial pressures
Hemodynamics | Baseline
  Pulmonary vascular resistance
Hemodynamics | At the end of each verticalization step (30th minute)
  Pulmonary vascular resistance
Hemodynamics | Baseline
  Pulmonary artery occlusion pressure
Hemodynamics | At the end of each verticalization step (30th minute)
  Pulmonary artery occlusion pressure
Hemodynamics | Baseline
  Systolic ejection volume
Hemodynamics | At the end of each verticalization step (30th minute)
  Systolic ejection volume
Hemodynamics | Baseline
  SvO2
Hemodynamics | At the end of each verticalization step (30th minute)
  SvO2
Hemodynamics | Baseline
  End-diastolic volume
Hemodynamics | At the end of each verticalization step (30th minute)
  End-diastolic volume
Hemodynamics | Baseline
  Systemic vascular resistance
Hemodynamics | At the end of each verticalization step (30th minute)
  Systemic vascular resistance
Hemodynamics | Baseline
  Right ventricular end-diastolic volume
Hemodynamics | At the end of each verticalization step (30th minute)
  Right ventricular end-diastolic volume
Hemodynamics | Baseline
  Right ventricular ejection fraction
Hemodynamics | At the end of each verticalization step (30th minute)
  Right ventricular ejection fraction
Blood gases | Baseline
  Arterial and mixed venous blood gases data (PaO2, PaCO2, SaO2, SvO2).
Blood gases | At the end of each verticalization step (30th minute)
  Arterial and mixed venous blood gases data (PaO2, PaCO2, SaO2, SvO2).

CONTACTS AND LOCATIONS:
Overall Officials: Jules Audard, Study Chair — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bouchant L, Godet T, Arpajou G, Aupetitgendre L, Cayot S, Guerin R, Jabaudon M, Verlhac C, Blondonnet R, Borao L, Pereira B, Constantin JM, Bazin JE, Futier E, Audard J. Physiological effects and safety of bed verticalization in patients with acute respiratory distress syndrome. Crit Care. 2024 Aug 5;28(1):262. doi: 10.1186/s13054-024-05013-y. PMID 39103928